CLINICAL TRIAL: NCT02037503
Title: Effects of Ketamine Treatment on Suicidal Ideation, Drug-resistant Major Depression, and Negative Emotional Experience. Clinical and fMRI Study
Brief Title: The Effect of Ketamine on Mechanises Underlying Suicidal Ideation and Drug-resistant Major Depression
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TASMC-13-TH-0270-CTIL
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2019-11

CONDITIONS: Suicidal Ideation; Major Depressive Disorder; Healthy Participants
MeSH Terms: conditions — Suicidal Ideation; Depressive Disorder, Major | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo for drug resistant depression (Placebo Comparator): Patients will be treated for 21 days with daily oral placebo
  Interventions: Drug: Saline
- Ketamine for suicidal ideation (Experimental): Patients will be treated for 21 days with daily oral Ketamine
  Interventions: Drug: Ketamine
- Ketamine for drug resistant depression (Experimental): Patients will be treated for 21 days with daily oral Ketamine
  Interventions: Drug: Ketamine
- Placebo in suicidal ideation (Placebo Comparator): Patients will be treated for 21 days with daily oral placebo
  Interventions: Drug: Saline
- Healthy Participants (Experimental): Healthy participants that underwent a romantic relationship breakup will attend in tow experimental sessions, one with placebo and one with ketamine. Sessions will be separated within the range of 1 to 6 weeks
  Interventions: Drug: Ketamine; Drug: Saline

INTERVENTIONS:
Drug: Ketamine
  Arms: Healthy Participants; Ketamine for drug resistant depression; Ketamine for suicidal ideation
Drug: Saline
  Arms: Healthy Participants; Placebo for drug resistant depression; Placebo in suicidal ideation

SUMMARY:
Suicide attempts are a serious concern worldwide. Currently, existing drugs take about three weeks to show effect on suicidal thoughts and drives. Recent evidence suggests that intravenous Ketamine exerts a rapid effect in suicidal patients, even after a single injection. We aim to examine whether oral Ketamine is a safe and effective treatment in suicidal patients. Following a suicide attempt, patients will be randomized into a group that will be given Ketamine for 21 days and one that will receive placebo, and assessed using questionnaires and brain scans. We expect early improvements in suicide scales in the Ketamine group.

As a secondary goal, this study will use IV ketamine in order to access the extent to which the experience of the embodied self mediate different levels of "embodied emotion". A better understanding of these relations will assist in unveiling the cognitive mechanism underlying the therapeutic effect of ketamine

DETAILED DESCRIPTION:
Suicide is a leading cause of death worldwide. Current strategies rely mostly on prevention, as there is no pharmacotherapy that seems to benefit patients in the acute phase of suicidal ideation. Conventional medications exert a beneficial effect only after three weeks. However, recent evidence suggests that intravenous Ketamine, an NMDA receptor antagonist, has a rapid and direct beneficial effect on suicidal ideation, even after a single dose.

We hypothesize that daily oral administration of Ketamine in suicidal patients will prove a safe and effective outpatient treatment.

In a double blind, placebo-controlled trial, patients admitted to the emergency department after a suicide attempt will be randomized into two groups: one will be given a daily sub-anesthetic dose of oral Ketamine, while the second group will receive a daily dose of placebo. Participants will be followed-up for 21 days. Some of the subjects will also undergo functional MRI scans before and after the first Ketamine intake.

We expect significant early improvements in suicide and depression scales in the active treatment group. If daily oral Ketamine proves a safe, cost-effective, and beneficial treatment option for suicidal ideation, this will constitute a much needed new tool in preventing suicide ideation related morbidity and mortality.

The secondary goal, delineating the relation between sense of embodied self and embodied emotion, will be approached by recruiting 40 healthy participants that underwent a romantic relationship break-up. Each participant will undergo two sessions: one under the placebo and the other under Ketamine. Each session will involve two main tasks: a virtual version of the rubber hand illusion and a task comparing mental and physical pain perception. The vRHI will involve four conditions that will be induced by two independent variables, synchronicity (synchronous-asynchronous) and pleasantness (high/low). The mental/physical pain task will include four conditions as well: Physical pain (high/low) and mental pain (high/low)

ELIGIBILITY:
Inclusion Criteria:

Suicidal Ideation group:

1. Any person admitted to the emergency room department after a suicide attempt , defined as requiring medical intervention - not just a psychiatrist ( surgical or pharmacological treatment but also the need for observation ) .
2. The need for medical intervention will be defined by the ER ED physician
3. Ages 18-65

For the depression group:

1. Diagnosed with major depression according to DSM VI.
2. Ongoing depression (according to DSM criteria) despite treatment with at least two antidepressants in adequate dosages and for longer than three weeks.
3. Ages 18-65

For the romantic relationship breakup:

1. Participants that have experienced a meaningful romantic relationship break-up within the past 12 months

-

Exclusion Criteria for all groups:

1. Psychotic state instate in the examination
2. Diagnosis of schizophrenia / schizoaffective disorder
3. Drug or alcohol abuse as is revealed in by blood/urine tests
4. Patient in which, according to the examiner, there is primary or secondary gain.
5. Patient , which, at the time of his admission , is without any pharmacological treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Resolution of suicidal ideation | within 3 weeks of enrolement

SECONDARY OUTCOMES:
Improvement in depression indices | within 3 weeks of treatment

OTHER OUTCOMES:
Study adherence | within 3 weeks after commencing treatment
  How many patients quit the study due to side effects of the medication
The visual analogue pain intensity scale | During the experiment session
  Reduction in subjective pain intensity

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, N/A = Not Applicable, Israel

REFERENCES:
- [Derived] Domany Y, Bleich-Cohen M, Tarrasch R, Meidan R, Litvak-Lazar O, Stoppleman N, Schreiber S, Bloch M, Hendler T, Sharon H. Repeated oral ketamine for out-patient treatment of resistant depression: randomised, double-blind, placebo-controlled, proof-of-concept study. Br J Psychiatry. 2019 Jan;214(1):20-26. doi: 10.1192/bjp.2018.196. Epub 2018 Sep 24. PMID 30246667